CLINICAL TRIAL: NCT07130032
Title: A Trial To Compare Efficacy And Safety Of Anti-PD-1/PD-L1 Antibodies In Combination With Bevacizumab And Metronomic Cyclophosphamide In Patients With Non-Small Cell Lung Cancer And Cutaneous Melanoma Previously Treated With Immune Checkpoint Blockade
Brief Title: Efficacy And Safety Of Anti-PD-1/PD-L1 Antibodies In Combination With Bevacizumab And Metronomic Cyclophosphamide In Patients With Non-Small Cell Lung Cancer And Cutaneous Melanoma Previously Treated With Immune Checkpoint Blockade
Acronym: reICB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EuroCityClinic LLC (Network)
Collaborators: First Pavlov State Medical University in St. Petersburg, Russia (Unknown)
Responsible Party: Principal Investigator, Aram Musaelyan, PhD, medical onсologist, EuroCityClinic LLC
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2025-08-14; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Non-small Cell Lung Cancer (NSCLC); Metastatic Cutaneous Melanoma
Keywords: Metastatic non-small cell lung cancer; Metastatic cutaneous melanoma; Immune checkpoint inhibitor; Bevacizumab; Metronomic cyclophosphamide
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NSCLC (n=60) (Experimental): The cohort of individuals with metastatic NSCLC will be treated with the reICB regimen (anti-PD(L)-1 antibodies+ cyclophosphamide+ bevacizumab) until disease progression or unacceptable toxicity.
  Interventions: Combination Product: reICB regimen (NSCLC)
- melanoma (n=30) (Experimental): The cohort of individuals with metastatic cutaneous melanoma will be treated with the reICB regimen (anti-PD(L)-1 antibodies+ cyclophosphamide+ bevacizumab) until disease progression or unacceptable toxicity.
  Interventions: Combination Product: reICB regimen (melanoma)

INTERVENTIONS:
Combination Product: reICB regimen (NSCLC) — * ICI (one of the following): Atezolizumab 1200 mg every 3 weeks/Nivolumab 240 mg every 2 weeks/Pembrolizumab 200 mg every 3 weeks
  * Cyclophosphamide 50 mg PO daily
  * Bevacizumab 7.5 mg/kg every 3 weeks
  Arms: NSCLC (n=60)
Combination Product: reICB regimen (melanoma) — * ICI (one of the following): Nivolumab 240 mg every 2 weeks/Pembrolizumab 200 mg every 3 weeks
  * Cyclophosphamide 50 mg PO daily
  * Bevacizumab 7.5 mg/kg every 3 weeks
  Arms: melanoma (n=30)

SUMMARY:
This study will evaluate efficacy and safety of anti-PD-1/PD-L1 antibodies combined with bevacizumab and metronomic cyclophosphamide in patients with metastatic non-small cell lung cancer (NSCLC) and cutaneous melanoma previously treated with immune checkpoint blockade (ICB). The hypotheses of this study are that a combination of ICB, cyclophosphamide, and bevacizumab prolongs progression-free survival and overall survival, and also increases rates of objective responses and disease control.

DETAILED DESCRIPTION:
The main challenge in treating metastatic non-small cell lung cancer (NSCLC) and cutaneous melanoma is acquired resistance to PD-1/PD-L1 blockade. Mechanisms of resistance include loss of antigen expression, defects in the IFN-γ signaling pathway, decreased PD-L1 expression, and upregulation of alternative immune checkpoints. Additionally, changes in the tumor microenvironment, such as an increase in regulatory T cells (Tregs), myeloid-derived suppressor cells, and angiogenesis, create an immunosuppressive environment that reduces T-cell activity.

Bevacizumab, a monoclonal antibody against VEGF-A, has demonstrated the ability to "normalize" tumor vasculature, thereby improving perfusion, reducing hypoxia, and facilitating immune cell infiltration into tumors. Results from several phase III trials in renal cell carcinoma, NSCLC, and hepatocellular carcinoma have shown that combining PD-1/PD-L1 antibodies with anti-VEGF therapy significantly improves ORR and progression-free survival (PFS) compared to using either immunotherapy alone or standard chemotherapy.

Metronomic chemotherapy involves administering low doses of cytotoxic agents continuously. This therapy targets tumor endothelial cells and modulates the immune milieu rather than direct cytotoxic elimination of malignant cells. Metronomic cyclophosphamide specifically depletes cells and activates effector cells. Additionally, metronomic cyclophosphamide can boost antigen presentation by activating dendritic cells, enhancing anti-tumor T-cell responses. In preclinical NSCLC models, combining metronomic cyclophosphamide with PD-1 blockade led to lasting tumor regression. This was due to the antiangiogenic and immunomodulatory properties of metronomic cyclophosphamide, resulting in reduced microvessel density and increased CD8⁺ T-cell infiltration.

Targeting multiple pathways of acquired resistance simultaneously with three agents can result in synergistic effects. This approach can convert immunologically "cold" tumors into "hot" ones. In preclinical studies, combining PD-L1 blockade with VEGF blockade increased T-cell infiltration and remodeled the vasculature, while combining PD-L1 blockade with metronomic chemotherapy improved antigen presentation and increased the ratio of effector-to-regulatory T-cells. In our recent retrospective study of 43 patients with metastatic NSCLC previously treated with ICIs, the safety and efficacy of rechallenging with ICIs and metronomic cyclophosphamide with or without bevacizumab were evaluated. The combination of ICIs with cyclophosphamide produced an ORR of 16.7%, a DCR of 75.0%, a median PFS of 5.8 months, and an OS of 15.4 months. In the cohort receiving oral cyclophosphamide plus bevacizumab, the ORR was 26.3%, DCR 78.9%, PFS 6.8 months, and OS 17.6 months. Adverse events related to treatment did not lead to discontinuation of the investigational therapy in either group.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Provide written informed consent
* Age ≥ 18 years
* Histologically confirmed diagnosis of NSCLC and cutaneous melanoma with distant metastases.
* No mutations in the EGFR gene, ALK, ROS1, RET gene translocations (in case of NSCLC).
* For NSCLC: the individuals had previously received anti-PD-(L)1 antibodies in combination with platinum-containing chemotherapy either in the first line or sequentially in the first and second lines for the treatment of metastatic disease.
* For NSCLC: the individuals had previously received anti-PD-(L)1 antibodies for >6 months and experienced disease progression.
* For cutaneous melanoma: the individuals had previously received anti-PD-1 antibodies either in combination with or without anti-CTLA4 therapy for metastatic disease. If the patient had the BRAF V600 mutation, they were also treated with BRAF and MEK inhibitors.
* For cutaneous melanoma: the patient has previously received anti-PD-1 antibodies with or without anti-CTLA4 therapy for metastatic disease for >6 months and experienced disease progression

Exclusion Criteria:

* Presence of clinically significant cardiovascular disease: severe or unstable ischemic heart disease, history of myocardial infarction, New York Heart Association Class III/IV congestive heart failure, ventricular arrhythmias.
* Stroke and/or transient ischemic attack within 6 months prior to screening;
* Uncontrolled hypertension
* History of previous malignancies except non-melanoma skin cancers, or in situ cervical or breast cancer unless a complete remission was achieved at least 2 years prior to randomization AND no additional therapy is required during the study period. Patients having hepatic involvement of cancer should be excluded as per investigator assessment.
* Patients with CNS metastases are eligible only if the metastases are adequately treated.
* Absolute neutrophil count (ANC) <1.5×109/L, platelet count <100×109/L, or hemoglobin <9.0 g/dL.
* Serum total bilirubin >1.5 × the upper limit of normal (ULN). Participants with Gilbert syndrome, bilirubin <2 X ULN, and normal AST/ALT are eligible;
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × ULN;
* Serum creatinine >1.5 × ULN.
* History of a thromboembolic event
* Presence of any allergic reactions to components of the study drugs
* Concomitant medications with a known risk of causing QT prolongation and/or Torsades de Pointes.
* Any parallel anti-cancer systemic therapy, radiation therapy
* Women who are pregnant or lactating;
* Presence of unresolved adverse events of grade 2 or higher toxicity, according to CTCAE v5.0 criteria, from prior therapy (except for alopecia or neurotoxicity grade≤2).
* Any other serious or uncontrolled medical disorder, active infection, physical examination finding, laboratory finding, altered mental status, or psychiatric condition that, in the opinion of the investigator, would limit a patient's ability to comply with the study requirements, substantially increase risk to the patient, or impact the interpretability of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2025-08-14 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Per immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) | From randomization until the first documentation of best overall response (up to 24 months)
  objective response rate (ORR) was defined as the proportion of participants whose best overall outcome included a confirmed complete response (CR) or partial response (PR). PR corresponds to a minimum 30% reduction in the total diameter of target lesions compared to the baseline measurements. CR indicates the total disappearance of all identified target lesions. Additionally, any pathological lymph nodes (classified as target or non-target) must shrink to a short axis measurement below 10 millimeters (mm).
Progression-free Survival (PFS) Per immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) | From randomization until the first documentation of objective progression or death, whichever comes first (up to 24 months)
  Progression-free survival (PFS) was defined as the time from randomization to the initial occurrence of documented disease progression (PD) or death from any cause, whichever occurs earlier. PD was characterized by at least a 20% enlargement in the total diameter of target lesions compared to the smallest sum recorded during the study, along with an absolute increase of 5 mm or more. The development of any new lesions was also classified as PD.
Overall Survival (OS) | From randomization until the first documentation of objective progression or death, whichever comes first (up to 24 months)
  Overall survival (OS) was measured as the duration (in months) from date of randomization to death resulting from any cause. Participants who had not experienced death by the time of data analysis were censored at their most recent confirmed date of survival.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) Per immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) | From randomization until the first documentation of objective progression or death, whichever comes first (up to 24 months)
  DCR defined as the proportion of participants with confirmed complete response (CR), partial response (PR), or stable disease (SD) as their best overall response. PR: A reduction of at least 30% in the total diameter of target lesions relative to the initial baseline measurements. CR: The complete resolution of all identified target lesions. Pathological lymph nodes (target or non-target) must also exhibit a short axis reduction to under 10 mm. SD: Lesions showing neither sufficient shrinkage to meet PR criteria nor sufficient growth to qualify as progressive disease (PD), using the smallest total lesion size recorded during the study as the reference point. PD: Defined as a minimum 20% increase in the total diameter of target lesions compared to the lowest recorded measurement (nadir), which must also include an absolute increase of ≥5 mm. The emergence of new lesions also constitutes PD.
Duration of Response (DOR) Per immune-related Response Evaluation Criteria in Solid Tumors (iRECIST) | From randomization until the first documentation of objective progression or death, whichever comes first (up to 24 months)
  DOR was measured as the time (in months) from the initial documentation of a partial response (PR) or complete response (CR) until the first confirmed instance of disease progression (PD) or death from any cause, whichever occurred earlier.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs | From start of study drug administration up to approximately 38 months
  An adverse event (AE) refers to any unfavorable or unintended medical event experienced by a participant in a clinical trial involving a medicinal product, regardless of whether it is causally linked to the treatment. A treatment-emergent adverse event (TEAE) was defined as an AE that: began on or after the start of treatment, had an unspecified onset date, existed prior to treatment but worsened in severity after treatment initiation, continuing until 30 days after the final dose of the study drug or the start of subsequent anti-tumor therapy (whichever occurred first). Additionally, serious adverse events (SAEs) deemed treatment-related were classified as TEAEs even if they occurred after this 30-day period. AEs with missing or unreported onset dates were also categorized as TEAEs. Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V. Orlov, Professor, Principal Investigator — EuroCityClinic LLC
Locations (1):
- EuroCityClinic LLC, Saint Petersburg, Sankt-Peterburg, Russia

IPD SHARING:
Plan to Share IPD: Yes